CLINICAL TRIAL: NCT02114125
Title: The Effects of Physical Activity and Cognitive Training in Improving Cognitive Function of Institutionalized Older Residents
Brief Title: Effects of the Physical Activity and Cognitive Training Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 201112011RID
Record Dates: First submitted 2012-11-02; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Cognitive Decline
Keywords: Physical activity; Cognitive training
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity | interventions — Exercise; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Usual Care Group: (No Intervention): Usual care consists of standard institutionalized services provided by physicians, nurses, and support staff (e.g., nurse assistants, social workers) in long-term care facilities.
- High-intensity physical activity (5PA) (Experimental): The intervention conducts the group-based physical activity, 5 days per- week for 8 weeks.
  Interventions: Behavioral: Physical Activity
- Low-intensity PA and CT(3PA+2CT) (Experimental): The intervention conducts 3 days per-week physical activity and 2 days per-week cognitive training for 8 weeks.
  Interventions: Behavioral: Physical Activity; Behavioral: Cognitive Training
- High-intensity PA and CT (5PA+5CT) (Experimental): The intervention conducts the individual-based, multi-domains cognitive training, 5days per- week and group-based physical activity, 5 days per- week and for 8 weeks.
  Interventions: Behavioral: Physical Activity; Behavioral: Cognitive Training
- Low-intensity cognitive training (2CT) (Experimental): The intervention conducts the individual-based, multi-domains cognitive training, 2 days per- week for 8 weeks.
  Interventions: Behavioral: Cognitive Training
- High-intensity cognitive training (5CT) (Experimental): The intervention conducts the individual-based, multi-domains cognitive training, 5 days per- week for 8 weeks.
  Interventions: Behavioral: Cognitive Training

INTERVENTIONS:
Behavioral: Physical Activity — group-based physical activity
  Arms: High-intensity PA and CT (5PA+5CT); High-intensity physical activity (5PA); Low-intensity PA and CT(3PA+2CT)
Behavioral: Cognitive Training — individual-based, multi-domains cognitive training
  Arms: High-intensity PA and CT (5PA+5CT); High-intensity cognitive training (5CT); Low-intensity PA and CT(3PA+2CT); Low-intensity cognitive training (2CT)

SUMMARY:
Investigators assume that there are some positive effects of cognitive training and physical activities on cognitive function, depression and quality of life in a sample of older residents in long-term care facilities.

The purpose of this study is to explore the effects of various interventions (physical activity, cognitive training, integration of physical activity and cognitive training) on different outcome indictors in institutionalized older residents.

DETAILED DESCRIPTION:
1. to develop an intervention protocol that achieves clinical development objectives in a scientifically rigorous and time efficient manner.
2. to further analyze the effects of the various interventions and make a comparison of dose-response relation and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 year and older
* Able to communicate verbally
* Able to discern 5*5 cm2 picture from a viewing distance of 20 cm
* Able to hear a sound of normal speech from a distance of 20 cm
* Able to sit in a chair or wheelchair independently for more than 30 minutes without changes in vital signs and awareness and without physical discomfort
* Has cognitive decline status assessing by CASI 2.0
* Lived in long-term care facilities during the study

Exclusion Criteria:

* Complete aphasia, blindness, deafness or completely dependent
* Unstable angina, arrythmia, myocardial infarction history, postural hypotension, transient cerebral hypoxia or other psychiatric disorders except depression
* Thrombophlebitis, or malignancy of the limbs.
* Refusal by patient or family member.
* Others. Reason to be well documented.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Cognitive Function at 8 weeks and 16weeks | pre-treatment (0 week, T0), post-treatment (8 weeks, T1) and follow-up (16 weeks, T2 )
  Cognitive Function: Cognitive Assessment Screening Instrument (CASI) 2.0 in Chinese version

SECONDARY OUTCOMES:
Change from Baseline Depression at 8 weeks and 16weeks | pre-treatment (0 week, T0), post-treatment (8 weeks, T1) and follow-up (16 weeks, T2 )
  Depression: Geriatric depression scale (GDS)-15 in Chinese version.
Change from Baseline Quality of Life at 8 weeks and 16weeksStatus: | pre-treatment (0 week, T0), post-treatment (8 weeks, T1) and follow-up (16 weeks, T2 )
  Quality of Life: Short Form-12 (SF-12) in Chinese version.

CONTACTS AND LOCATIONS:
Overall Officials: Meei-Fang Lou, PhD, Principal Investigator — Department of Nursing, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan Unversity Hospital, Taipei, Taiwan, Taiwan